CLINICAL TRIAL: NCT02092688
Title: Evaluation of a Novel Diagnostic Kit for the Detection of Placental Alpha-Microglobulin-1 in the Prediction of Preterm Birth in Women Presenting With Signs and Symptoms of Preterm Labor in Comparison to a Control Group of Asymptomatic Women With the Same Gestational Age - a Multicenter Trial
Brief Title: Evaluation of a Novel Diagnostic Kit for the Detection of Placental Alpha-Microglobulin-1 in the Prediction of Preterm Birth
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: AmniSure International LLC (Other)
Responsible Party: Sponsor
Other Study IDs: 140/13
Record Dates: First submitted 2014-02-26; First posted 2014-03-20 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Preterm Labour; Preterm Birth
Keywords: time to delivery; PROM; PTL; positive predictive value
MeSH Terms: conditions — Obstetric Labor, Premature; Premature Birth

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Study group: Study group: women between 24 and 36 6/7 weeks of gestation that present with self-reported signs, symptoms or complaints suggestive of preterm labor
  Interventions: Device: novel kit for the detection of PAMG-1
- Control group: Control group: women between 24 and 36 6/7 weeks of gestation without signs or symptoms of PTL
  Interventions: Device: novel kit for the detection of PAMG-1

INTERVENTIONS:
Device: novel kit for the detection of PAMG-1 — The novel kit for the detection of PAMG-1 is a diagnostic device employing monoclonal antibodies that detect Placental α1 Microglobulin present in cervico-vaginal secretions manufactured by AmniSure® International, LLC, Boston, MA. The in vivo sensitivity detection threshold is 4ng/ml. During the test procedure, PAMG-1 from the sample sequentially binds to monoclonal antibody conjugated with labeled particles, then to monoclonal antibody immobilized on an insoluble carrier. The test requires a 30 second swab saturation in the vagina (a sterile speculum examination is not required), a 30 second active washing step whereby the swab just removed from the vagina is actively rotated in a solvent filled vial and lastly, a 5 minute waiting period from the time the swab is removed and the test strip is inserted if two testing lines do not appear sooner.

SUMMARY:
This is a prospective observational trial that will enroll pregnant women between 24 and 36 6/7 weeks of gestation that present with signs and symptom of preterm labor with clinically intact membranes and cervical dilatation ≤ 3 cm and a control group of pregnant women without signs and risks for PTL to assess how the results of the novel kit for the detection of PAMG-1 in both patient groups correlate to their time-to-delivery (TTD) and other adverse neonatal and pregnancy outcomes.

Thes study hypothesis contains that the novel diagnostic kit will identify women who are at high risk for preterm birth by a high positive predictive value.

DETAILED DESCRIPTION:
Background

Placental alpha microglobulin-1 (PAMG-1) is a protein found in high concentrations in amniotic fluid but very low concentrations in background levels of cervico-vaginal discharge. In recent years, the medical community has increasingly accepted the widespread use of detecting PAMG-1 to aid the provider in confirming or ruling out rupture of the fetal membranes (ROM). The test used is commercially marketed as the AmniSure® ROM Test, manufactured by AmniSure® International, LLC, Boston, MA, USA.

In one of the original investigations of PAMG-1 for the detection of ROM, Lee et al. noted that in 20 out of the 23 cases where the AmniSure® ROM Test was positive and standard clinical assessment (i.e. nitrazine, ferning and pooling) was negative, the patient was ultimately determined to have been ruptured upon retrospective analysis of their clinical course. It was later reported that for all of the preterm patients in this group that showed signs and symptoms of labor, delivery followed within 7 days. In 2011, the clinical value of a positive AmniSure® ROM Test in the patient presenting with signs and symptoms of preterm labor (PTL) but without membrane rupture was investigated by this same group. The results demonstrated that the AmniSure® ROM Test was highly predictive of delivery of these patients within 48 hours, 7 days and 14 days.

In the patient group on whom the above tests are performed, membrane rupture is excluded as this condition, if present, confirms imminent delivery and dictates a different course of management. It has been demonstrated that the AmniSure® ROM Test can detect PAMG-1 in patients presenting with signs and symptoms of ROM when all other traditional methods are unable to do so. The likelihoods of adverse outcomes associated with these sub-clinical ruptures have been demonstrated to not be statistically different from the adverse outcomes associated with gross or clinically detectable ruptures. The proposed physiological explanation for this phenomenon is that PAMG-1 is released through micro-perforations of the amniotic membranes that more copious amounts of fluid cannot pass through.

The major difference, however, between the patient presenting with signs of preterm labor and those just described above is the presence, or absence, of membrane rupture signs or complaints. Given that the complaints of ROM are typically rooted in an overt episode of suspicious fluid leakage, it is hypothesized that the resulting concentration of PAMG-1 in the vagina of the patient without such overt complaints or signs of ROM will be lower than the current sensitivity threshold of the AmniSure® ROM Test.

Accordingly, a device that is more sensitive in its detection of PAMG-1 than the AmniSure® ROM Test presumably will be able to detect more patients at risk for imminent delivery than its predecessor in patients presenting to labor and delivery units with signs, symptoms or complaints suggestive of preterm labor (PTL) who have no clinical evidence of membrane rupture. If this is the case, this tool may be of significant value to the provider in deciding how to manage their patients suspected to be at risk for imminent delivery. Management options may include administration of tocolytics to prolong gestation, corticosteroids to improve respiratory development, administration of antibiotics to decrease the risk of infection (intra-partum and post-partum), prescription of bed rest, as well as increased observation and fetal monitoring.

Currently, the American College of Obstetricians and Gynecologists (ACOG) indicate in their most recent Practice Bulletin on the Management of Preterm Labor that many tests to identify women at risk of preterm birth have been proposed and evaluated; however, only ultrasonography and fetal fibronectin testing have been shown to have benefit. Ultrasonography to determine cervical length, fetal fibronectin testing, or a combination of both may be useful in determining which women are at high risk for preterm delivery. However, their clinical usefulness may rest primarily with their ability to identify women who are least likely to deliver (i.e. their negative predictive value). Therefore, there is an urgent need for a test with a high positive predictive value in order to accurately predict imminent delivery to allow for salutary intervention.

Objective

1. To assess the efficacy of the novel kit for the detection of PAMG-1 in the cervico-vaginal secretions of pregnant women with clinically intact membranes presenting with signs and symptoms of PTL in predicting time-to-delivery. Assessment will be stratified by the following gestational age ranges:

   1. 24-31 6/7 weeks
   2. 32-36 6/7 weeks
2. To compare the results of the novel kit for the detection of PAMG-1 in pregnant women presenting with signs of PTL to a control group of pregnant women with the same gestational age without any symptoms and without an elevated risk of preterm birth.
3. To compare the novel kit for the detection of PAMG-1 to other methods available in assessing time to delivery in the same patient population, including:

   1. cervical length measurements by trans-vaginal ultrasound
   2. cervical dilatation > 1 cm
   3. Contraction Frequency ≥ 6 per hour (one every 10 min)
4. Determine the association between the results of the kit, cervical length and neonatal outcomes.

Methods

1. Study group: Patient presenting with symptoms of PTL between 24 and 36 6/7 weeks of gestation signs informed consent.

   Control group: Patient presenting for routine pregnancy control without any symptoms of PTL is between 24 an 36 6/7 weeks of gestation signs informed consent.
2. Specimen for the PAMG-1 test is collected in accordance with manufacturer's recommendations. During the same examination the physician takes a vaginal microbiological smear.
3. The sample is labeled and stored for later examination by a separate investigator who will not know the results of the physician's regular clinical evaluation.
4. After the physician completes their physical examination of the patient.
5. Cervical length measurement by transvaginal ultrasound (TVU) is performed.
6. Patient delivery data (e.g. time, condition, etc.) are recorded in the follow up.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting for emergency obstetrical care at an emergency room or labor & delivery unit with signs, symptoms or complaints suggestive of preterm labor (PTL)
* Gestational age between 24 and 36 6/7 weeks of gestation
* Consenting to be part of the trial
* Women between 24 and 36 6/7 weeks of gestation without signs or symptoms of PTL
* Written informed consent

Exclusion Criteria

* PROM
* > 3 cm cervical dilatation
* < 18 yrs old and not emancipated consenting minor
* Heavy vaginal bleeding
* Cervical dilatation > 3 centimeters
* Suspected placenta previa
* < 24 weeks of gestation or ≥ 37 weeks of gestation
* Cervical cerclage in place or cervical pessary
* A symptom not associated with idiopathic threatened preterm delivery (e.g. trauma)
* Enrollment in a tocolytic study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: pregnant women presenting with signs auf PTL at emergenca care and pregnant asymptomatic women presenting for routine check-up
Sampling Method: Non-Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2013-12; Primary Completion 2016-12-31 (Actual); Study Completion 2017-03-31 (Actual)

PRIMARY OUTCOMES:
Time to delivery | 3 months
  Measured in days

SECONDARY OUTCOMES:
Number of patients who have a positive PAMG-1-Test and deliver within 48 hours, 7 days and 14 days after taking the test | 3 months
Number of patients who have a negative PAMG-1-Test and do not deliver within 48 hours, 7 days and 14 days after taking the test | 3 months
Time of delivery | 37 weeks
  Measured in weeks
Number of babies admitted to NICU | 3 months
Number of babies with histological chorioamnionitis | 3 months
Number of babies with respiratory distress syndrome | 3 months
Time to Delivery | 3 months
  Measured in weeks; prolongation of delivery from administration
Number of babies with infection | 3 months
Number of babies with intracranial hemorrhage | 3 months
Number of babies with necrotizing enterocolitis | 3 months
Number of babies with patent ductus arteriosus | 3 months
Number of babies with neonatal sepsis | 3 months
Birthweight | 3 months
  Measured in grams
Number of perinatal deaths | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Surbek, Prof. Dr. med., Principal Investigator — Geburtshilfe Frauenklinik Inselspital
Locations (1):
- Prof. Dr. Daniel Surbek, Bern, Switzerland

REFERENCES:
- [Background] Di Renzo GC, Roura LC, Facchinetti F, Antsaklis A, Breborowicz G, Gratacos E, Husslein P, Lamont R, Mikhailov A, Montenegro N, Radunovic N, Robson M, Robson SC, Sen C, Shennan A, Stamatian F, Ville Y. Guidelines for the management of spontaneous preterm labor: identification of spontaneous preterm labor, diagnosis of preterm premature rupture of membranes, and preventive tools for preterm birth. J Matern Fetal Neonatal Med. 2011 May;24(5):659-67. doi: 10.3109/14767058.2011.553694. Epub 2011 Mar 2. No abstract available. PMID 21366393
- [Background] Gungorduk K, Asicioglu O, Besimoglu B, Gungorduk OC, Yildirm G, Ark C, Sahbaz A. Labor induction in term premature rupture of membranes: comparison between oxytocin and dinoprostone followed 6 hours later by oxytocin. Am J Obstet Gynecol. 2012 Jan;206(1):60.e1-8. doi: 10.1016/j.ajog.2011.07.035. Epub 2011 Jul 30. PMID 21924396
- [Background] Kurdoglu M, Kolusari A, Adali E, Yildizhan R, Kurdoglu Z, Kucukaydin Z, Kaya A, Kirimi E, Sahin HG, Kamaci M. Does residual amniotic fluid after preterm premature rupture of membranes have an effect on perinatal outcomes? 12 years experience of a tertiary care center. Arch Gynecol Obstet. 2010 Apr;281(4):601-7. doi: 10.1007/s00404-009-1147-4. Epub 2009 Jun 12. PMID 19521709
- [Background] Lee SE, Park JS, Norwitz ER, Kim KW, Park HS, Jun JK. Measurement of placental alpha-microglobulin-1 in cervicovaginal discharge to diagnose rupture of membranes. Obstet Gynecol. 2007 Mar;109(3):634-40. doi: 10.1097/01.AOG.0000252706.46734.0a. PMID 17329514
- [Background] Lee SM, Lee J, Seong HS, Lee SE, Park JS, Romero R, Yoon BH. The clinical significance of a positive Amnisure test in women with term labor with intact membranes. J Matern Fetal Neonatal Med. 2009 Apr;22(4):305-10. doi: 10.1080/14767050902801694. PMID 19350444
- [Background] Lee SM, Romero R, Park JW, Kim SM, Park CW, Korzeniewski SJ, Chaiworapongsa T, Yoon BH. The clinical significance of a positive Amnisure test in women with preterm labor and intact membranes. J Matern Fetal Neonatal Med. 2012 Sep;25(9):1690-8. doi: 10.3109/14767058.2012.657279. Epub 2012 Apr 25. PMID 22280400